CLINICAL TRIAL: NCT02593162
Title: Phase 2a, Randomized, Double-Blind Study to Investigate the Safety and Efficacy of Faldaprevir in Combination With Ribavirin and TD-6450 for 12 Weeks in Treatment-Naive Patients Chronically Infected With Genotype 4 Hepatitis C Virus
Brief Title: A Study of Faldaprevir, Ribavirin and TD-6450 in Participants With Genotype 4 Hepatitis C Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trek Therapeutics, PBC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRK-450-0201
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Hepatitis C Viral Infection; Chronic Hepatitis C; Hepatitis C (HCV); Hepatitis C Genotype 4
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — faldaprevir; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): 12 weeks of Faldaprevir plus low dose TD-6450 plus Ribavirin
  Interventions: Drug: Faldaprevir; Drug: TD-6450; Drug: Ribavirin
- Group 2 (Experimental): 12 weeks of Faldaprevir plus high dose TD-6450 plus Ribavirin
  Interventions: Drug: Faldaprevir; Drug: TD-6450; Drug: Ribavirin

INTERVENTIONS:
Drug: Faldaprevir
  Other Names: BI 201335
Drug: TD-6450
Drug: Ribavirin
  Other Names: Ribasphere®

SUMMARY:
Phase 2a study designed to assess the safety, efficacy, and pharmacokinetics of Faldaprevir and TD-6450 in combination with Ribavirin for a 12-week treatment duration in treatment-naïve participants with genotype 4 hepatitis C virus (HCV) infection.

DETAILED DESCRIPTION:
A study to evaluate the safety and effect of treatment with experimental antiviral drugs in combination with ribavirin in treatment-naïve participants with genotype 4 hepatitis C infection. The study will test the safety and effects of this alternative treatment for up to 12 weeks. Secondary objectives of this study are to determine the pharmacokinetics of the study drugs when co-administered, and to evaluate HCV RNA kinetics during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic genotype 4 hepatitis C infection and HCV RNA ≥ 10^4 IU/mL at screening
* Hepatitis C virus treatment naive, defined as defined as having never received a direct acting anti-viral (DAA), and as having received ≤ 8 weeks of interferon ≥ 6 months prior to screening
* Absence of cirrhosis as defined by one of the following:

  * A liver biopsy performed within 24 calendar months of Day 1 showing absence of cirrhosis
  * Transient elastography (FibroScan®) performed within 12 calendar months of Day 1 with a result of ≤ 12.5 kPa
  * A FibroSure® score ≤ 0.48 and AST:platelet ratio (APRI) ≤ 1 performed during screening

Exclusion Criteria:

* Infection with hepatitis B virus (HBV) or human immunodeficiency virus, HIV-1 or HIV-2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving 12-week sustained virologic response following treatment with 2 direct acting anti-virals and ribavirin in Genotype 4 Hepatitis C infected adults | Post Treatment Week 12

SECONDARY OUTCOMES:
Percentage of subjects with virologic response at Week 12 (HCV RNA less than lower limit of quantitation at end of therapy with Faldaprevir plus TD-6450 plus ribavirin) | Week 12
Percentage of subjects with virologic response 2, 4 and 8 weeks after treatment completion (HCV RNA less than lower limit of quantitation at 2, 4 and 8 weeks after end of therapy with Faldaprevir plus TD-6450 plus ribavirin) | Post Treatment Weeks 2 to 8

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Hassanein, MD, Principal Investigator — Southern California Research Center
Locations (1):
- Southern California Research Center, Coronado, California, United States

IPD SHARING:
Plan to Share IPD: No